CLINICAL TRIAL: NCT01668264
Title: Combined Echocardiographic and MRI Assessment of Diastolic Function in Patients With Congenital Heart Disease
Brief Title: Imaging Assessment of Diastolic Function
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Luc Mertens, Staff Cardiologist, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000017963
Record Dates: First submitted 2012-08-13; First posted 2012-08-20 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Congenital Heart Disease
Keywords: Pediatrics; Congenital Heart Disease; Diastolic Function; Echocardiograph; MRI
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnetic Resonance Imaging (MRI) (Experimental): Subjects with congenital heart disease will undergo an echocardiograph, as well as an MRI.
  Interventions: Procedure: Echocardiograph; Procedure: Magnetic Resonance Imaging (MRI)
- Echocardiograph (Experimental): Subjects with congenital heart disease will undergo an echocardiograph, as well as an MRI.
  Interventions: Procedure: Echocardiograph; Procedure: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Procedure: Echocardiograph
Procedure: Magnetic Resonance Imaging (MRI)

SUMMARY:
Diastolic function is poorly studied in children with congenital heart disease. This is mainly due to the lack of validated techniques. Cardiac MRI offers two advantages compared to echocardiography: 1. accurate measurements of ventricular volumes and mass; 2. tissue characterization. The main advantage of echocardiography is a better temporal resolution which allows the study of short events like early relaxation. Overall there is a lack of studies correlating different echocardiographic and MRI parameters of heart function in pediatric populations with congenital or acquired heart diseases. This study will address specific questions on specific groups of patients that might bring more insight into chamber interaction and cardiac function. This study hypothesizes the following:

* Atrial enlargement is a marker of chronic increase in filling pressures and 3D echo might be the best method for follow-up.
* Cardiac remodeling associated with chronic loading results in changes in diastolic properties related to changes in cardiac mass and volume. This is related to changes in cardiac mechanics influencing diastolic parameters. Especially the influence on twisting and untwisting will be studied.
* Regional myocardial fibrosis and scarring may account for regional systolic and diastolic dysfunction with possible prognostic impact

ELIGIBILITY:
Inclusion Criteria:

* All patients with tetralogy of Fallot post repair, transposition of great arteries after arterial switch operation, aortic valvulopathy (aortic stenosis and aortic regurgitation), coarctation of the aorta and cardiomyopathy, who are planned to undergo a cardiac MRI will be eligible.
* Informed consent

Exclusion Criteria:

* Lack of informed consent
* Need for general anesthesia
* Similar contraindications as for a clinical MRI study apply.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)

PRIMARY OUTCOMES:
Atrial Volumes | Day 1
  Measure right and left atrial volumes by 2D and 3D echo and correlate the different echocardiographic measurements with MRI. This will allow identifying the most accurate measurement which can be used in clinical practice.

SECONDARY OUTCOMES:
Assess Ventricular Volumes | Day 1
  Assess ventricular volumes and mass and calculate mass/volume ratio. Study the effect of ventricular remodeling on myocardial mechanics especially twisting and untwisting. Relate these changes to evaluation of diastolic function.
Myocardial Scarring | Day 1
  Assess the presence of myocardial scarring in specific populations with congenital heart disease and correlate the findings with regional and global systolic and diastolic dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Mertens, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada